CLINICAL TRIAL: NCT07220980
Title: Optimal Duration of Indwelling Urethral Foley Catheter Following Bulbar Urethroplasty: A Pragmatic Multi-Institutional Randomized Controlled Non-Inferiority Trial
Brief Title: Optimal Duration of Foley Catheter After Bulbar Urethroplasty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jane Kurtzman (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Jane Kurtzman, Assistant Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 171398
Record Dates: First submitted 2025-10-22; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Urethral Stricture, Bulbar
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Early Removal (Experimental)
  Interventions: Device: Early catheter removal
- Later Removal (Experimental)
  Interventions: Device: Later catheter removal

INTERVENTIONS:
Device: Early catheter removal — Removal after 7-10 days
  Arms: Early Removal
Device: Later catheter removal — Removal after 18-21 days
  Arms: Later Removal

SUMMARY:
The goal of this clinical trial is to learn when is the best time to remove a Foley catheter (tube used to drain urine from the bladder) after surgery in adult men who have a specific type of urethral stricture disease (narrowing of the tube that carries urine from the body). The main question it aims to answer is:

- Is there a difference between removing the catheter at 7-10 days versus 18-21 days?

Researchers will compare Foley removal at 7-10 days to removal at 18-21 days to see if there is a difference in problems after surgery or if the narrowing returns.

Participants will:

* Complete a survey before surgery, when the catheter is removed, and within 12 months after surgery
* Complete follow-up visits after surgery based on your specific medical needs and standard of care

ELIGIBILITY:
Inclusion Criteria:

* Cis-male patients
* Age 18-70, inclusive
* Bulbar urethral stricture undergoing a urethroplasty
* Urethral stricture defect less than or equal to 7cm in length
* First time urethroplasty
* Negative urine analysis or urine culture

Exclusion Criteria:

* History of pelvic radiation
* Diabetes with Hba1c greater than 8%
* Penile urethral stricture
* Posterior urethroplasty
* Bulbar stricture greater than 7cm

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience a Stricture Recurrence | 1 year
Number of Participants who Experience a Perioperative Complication | From Foley insertion to Foley removal

SECONDARY OUTCOMES:
Rate of Retrograde Urethrograms Performed on Day of Foley Removal | Foley Removal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No